CLINICAL TRIAL: NCT03883919
Title: A Pilot Study of Liposomal Irinotecan Plus 5-FU / LV Combined With Paricalcitol in Patients With Advanced Pancreatic Cancer Progressed on Gemcitabine-based Therapy
Brief Title: Liposomal Irinotecan Plus 5-FU / LV Combined With Paricalcitol in Patients With Advanced Pancreatic Cancer Progressed on Gemcitabine-based Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201905201
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer; Pancreas Cancer; Cancer of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Leucovorin; irinotecan sucrosofate; paricalcitol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Paricalcitol 75 mcg Days 1 and 8 (Experimental): * 5-FU, LV, and nal-IRI will be administered at standard fixed doses. Briefly, 5-FU will be given at a dose of 2400 mg/m^2 continuous IV infusion over 46 hours, LV will be given at 400 mg/m^2 IV over 30 minutes, and liposomal irinotecan will be given at a dose of 70 mg/m^2 IV over 90 minutes (unless homozygous for the UGT1A1*28 7/7 allele, in which case the dose will start at 50 mg/m^2 and escalate to 70 mg/m^2 in subsequent cycles if no excessive toxicity is experienced) on Day 1 of each 14-day cycle.
  * Paricalcitol 75 mcg on Days 1 and 8
  * Treatment with liposomal irinotecan plus 5FU/ LV may continue indefinitely, and treatment with paricalcitol may continue for up to 10 cycles (20 weeks)
  Interventions: Drug: 5-FU; Drug: Leucovorin; Drug: Liposomal Irinotecan; Drug: Paricalcitol; Procedure: Serum and plasma blood samples; Procedure: Tumor biopsy
- Group 2: Paricalcitol 7 mcg/kg Days 1 and 8 (Experimental): * 5-FU, LV, and nal-IRI will be administered at standard fixed doses. Briefly, 5-FU will be given at a dose of 2400 mg/m^2 continuous IV infusion over 46 hours, LV will be given at 400 mg/m^2 IV over 30 minutes, and liposomal irinotecan will be given at a dose of 70 mg/m^2 IV over 90 minutes (unless homozygous for the UGT1A1*28 7/7 allele, in which case the dose will start at 50 mg/m^2 and escalate to 70 mg/m^2 in subsequent cycles if no excessive toxicity is experienced) on Day 1 of each 14-day cycle.
  * Paricalcitol 7 mcg/kg on Days 1 and 8
  * Treatment with liposomal irinotecan plus 5FU/ LV may continue indefinitely, and treatment with paricalcitol may continue for up to 10 cycles (20 weeks)
  Interventions: Drug: 5-FU; Drug: Leucovorin; Drug: Liposomal Irinotecan; Drug: Paricalcitol; Procedure: Serum and plasma blood samples; Procedure: Tumor biopsy

INTERVENTIONS:
Drug: 5-FU — -Standard of care drug
  Other Names: Fluorouracil; Adrucil
Drug: Leucovorin — -Standard of care drug
  Other Names: Wellcovorin; Folinic acid
Drug: Liposomal Irinotecan — -Standard of care drug
  Other Names: nal-IRI; Onivyde
Drug: Paricalcitol — -Investigational drug
  Other Names: Zemplar; Vitamin D
Procedure: Serum and plasma blood samples — -baseline, day 1 of each cycle beginning with cycle 2
Procedure: Tumor biopsy — * 5 patients in each arm will be required to undergo a mandatory tumor biopsy from the primary pancreatic site or metastatic site, if safe and feasible, prior to cycle 1
  * After Cycle 3 of treatment, all patients who had a baseline biopsy will be required to undergo a mandatory biopsy of the same site if safe and feasible.

SUMMARY:
Given the efficacy of nanoliposomal irinotecan as a second-line regimen in pancreatic ductal adenocarcinoma (PDAC), together with the favorable toxicity profile of paricalcitol and its interplay with irinotecan metabolism, the investigators propose a second-line pilot study in advanced PDAC that will enroll patients who have progressed on a gemcitabine-based regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma.
* Must have progressed on or become intolerant to gemcitabine-containing therapy in the advanced setting (not resectable). This is intended to be a second-line trial.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* At least 18 years of age.
* Life expectancy > 3 months.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 x ULN
  * Serum albumin > 3g/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN unless there are liver metastases, in which case AST and ALT ≤ 5.0 x IULN
  * Creatinine ≤ 1.5 x IULN OR GFR > 50 mL/min
  * Corrected calcium < 10.3 mg/dL
  * Phosphorus ≤ 4.5 mg/dL
* Patients will require a 2-week washout period from previous gemcitabine-based systemic therapy, a 2-week washout period from previous radiation therapy, and a 4-week washout period from major surgery prior to the first planned dose of study treatment.
* Prior clinically significant treatment-related toxicity must recover to grade 1 or less prior to the first planned dose of study treatment.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* More than one prior systemic treatment in the advanced setting. Disease recurrence within 6 months of adjuvant therapy is considered one line of systemic treatment.
* Patients with active renal, ureteral, or bladder stones on the screening imaging.
* Current use of or anticipated need for alternative, holistic, naturopathic, or botanical formulations used for the purpose of cancer treatment.
* A history of other malignancy within 2 years previous, with the exception of those basal cell or squamous cell carcinoma of the skin which were treated with local resection only, or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents.
* Patients who received FOLFIRINOX or FOLFIRI in the neoadjuvant or adjuvant setting who experienced disease recurrence within 6 months will be excluded (patients who received 5-FU or capecitabine as a radiosensitizer are permitted to enroll.)
* Patients with known active/ progressive brain metastases or leptomeningeal involvement will be excluded due to their poor prognosis. Patients with treated/stable brain metastases, defined as patients who have received prior therapy for their brain metastases and whose CNS disease is radiographically stable at study entry, are eligible.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to paricalcitol, liposomal irinotecan, 5-FU, LV, or other agents used in the study.
* Clinically significant ascites that requires therapeutic paracentesis or significant pleural effusion that requires therapeutic thoracentesis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of study entry.
* Known HIV-positivity not on anti-retroviral therapy, or with CD4+ T cell count < 200/ul (patients with known HIV currently on anti-retroviral therapy with CD4+ T cell count > 200/ul will be included).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Tolerability between two different dose levels of paricalcitol added to the combo regimen of liposomal irinotecan plus 5-FU / LV as measured by the occurrence of grade 3 and 4 toxicities | Through 30 days after completion of paricalcitol treatment (estimated to be 28 weeks)
  -Toxicity will be graded using CTCAE version 5.0

SECONDARY OUTCOMES:
Overall response rate (ORR) | Through completion of treatment (estimated to be 20 weeks)
  * The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 72 weeks)
  * PFS: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Overall survival (OS) | Through completion of follow-up (estimated to be 72 weeks)
  -Overall survival (OS) is defined as the date from treatment to death or last follow-up.
CA19-9 biochemical response rate | Through beginning of cycle 10 (estimated to be 18 weeks)
  -The biochemical response (BR) is defined as more than 50% of decrease from baseline CA 19-9.
Duration of overall response | Through completion of treatment (estimated to be 20 weeks)
  - The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Duration of complete response | Through completion of treatment (estimated to be 20 weeks)
  * The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and disappearance of all non-target lesions and normalization of tumor marker level.
Duration of stable disease | Through completion of treatment (estimated to be 20 weeks)
  * Duration of stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

CONTACTS AND LOCATIONS:
Overall Officials: Kian-Huat Lim, M.D, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan for sharing IPD to be determined.
Time Frame: Time frame for accessing IPD to be determined.
Access Criteria: Access criteria for sharing IPD to be determined.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu